CLINICAL TRIAL: NCT07065539
Title: The Impact of Duration of Gonadotropin-Releasing Hormone Agonist Pretreatment and Letrozole Supplementation on Pregnancy Outcomes in Frozen-Thawed Embryo Transfer Cycles for Patients With Adenomyosis: A 2 by 2 Factorial Multicenter, Randomized Controlled Trial
Brief Title: GnRH Agonist Pretreatment Duration and Letrozole Supplementation in Frozen Embryo Transfer for Adenomyosis Patients
Acronym: GOLD-FET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Women and Children's Hospital of Fujian Province (Unknown); BoAi Hospital of Zhongshan (Other)
Responsible Party: Principal Investigator, Yanwen Xu, Director of the Reproductive Medical Center, the First Affliated Hospital of Sun Yat-sen University, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2025012-5010
Record Dates: First submitted 2025-06-13; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Adenomyosis of Uterus; Frozen Embryo Transfer (FET)
Keywords: adenomyosis; embryo transfer; GnRH-a; letrozole; pre-treament
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- GnRH-a-1M (Active Comparator)
  Interventions: Drug: GnRH-a-1M
- GnRH-a-2M (Active Comparator)
  Interventions: Drug: GnRH-a-2M
- GnRH-a+LE-1M (Active Comparator)
  Interventions: Drug: GnRH-a+LE-1M
- GnRH-a+LE-2M (Active Comparator)
  Interventions: Drug: GnRH-a+LE-2M

INTERVENTIONS:
Drug: GnRH-a-1M — Pre-treatment with one dose GnRH agonist before endometrial preparation.
  Arms: GnRH-a-1M
Drug: GnRH-a-2M — Pre-treatment with two doses GnRH agonist before endometrial preparation.
  Arms: GnRH-a-2M
Drug: GnRH-a+LE-1M — Pre-treatment with one dose GnRH agonist, along with daily 2.5 mg letrozole for 28 days before endometrial preparation.
  Arms: GnRH-a+LE-1M
Drug: GnRH-a+LE-2M — Pre-treatment with two doses GnRH agonist, along with daily 2.5 mg letrozole for 28 days since the first injection of GnRH agonist before endometrial preparation.
  Arms: GnRH-a+LE-2M

SUMMARY:
This randomized clinical trial aims to assess the comparative effectiveness of different pre-treatment protocols prior to frozen embryo transfer (FET) among women with adenomyosis, providing evidence-based guidance for clinical decision-making. The main questions it aims to answer are:

Does the protocol involving two doses of gonadotropin-releasing hormone agonist (GnRH-a) pretreatment result in a higher live birth rate compared to one dose of GnRH-a pretreatment in women with adenomyosis undergoing frozen embryo transfer? Does the protocol involving GnRH-a with letrozole supplementation result in a higher live birth rate compared to GnRH-a monotherapy in women with adenomyosis undergoing frozen embryo transfer? Eligible participants will undergo screening before endometrial preparation for FET, following which they will be randomly assigned to one of four groups: GnRH-a-1M, GnRH-a-2M, GnRH-a+LE-1M or GnRH-a+LE-2M. In the GnRH-a-1M group, participants will be pre-treated with one dose GnRH agonist before endometrial preparation. In the GnRH-a-2M group, participants will be pre-treated with two doses GnRH agonist before endometrial preparation. In the GnRH-a+LE-1M group, participants will be pre-treated with one dose GnRH agonist and letrozole 28 days before endometrial preparation. In the GnRH-a+LE-2M group, participants will be pre-treated with two doses GnRH agonist, along with daily 2.5 mg letrozole for 28 days since the first injection of GnRH agonist before endometrial preparation. After pre-treament, all participants will return for endometrial preparation in artificial cycles.

ELIGIBILITY:
Inclusion Criteria:

* Sonographically diagnosed adenomyosis via transvaginal ultrasound;
* Candidates scheduled for frozen single blastocyst (Day5, Day6) transfer
* Age 20-38 years
* Previous embryo transfer attempts: ≤2 cycles

Exclusion Criteria:

* Patients diagnosed with Recurrent pregnancy loss, Autoimmune disorders (e.g., systemic lupus erythematosus), Uterine fibroids ≥5 cm, Cervical incompetence, Cesarean scar niche
* History of Myomectomy and/or adenomyosis lesion excision, Cervical conization
* Patients presenting with Congenital Müllerian anomalies (unicornuate uterus, septate uterus, etc.), Endometrial atypical hyperplasia, malignancy or defects
* Sperm retrieval method: Micro-TESE (microdissection testicular sperm extraction)
* Fertilization method: Rescue ICSI
* Endometrial thickness <7 mm, Intrauterine adhesions, Intrauterine fluid
* Contraindications to exogenous hormone administration
* Use of GnRH within 3 months prior to enrollment

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 432 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 40 weeks after embryo transfer

SECONDARY OUTCOMES:
Cycle Cancellation Rate | 3 weeks after initiating artificial cycle
Hypoestrogenic Adverse Event Rate | 4 weeks after 3.75mg GnRH-a intramuscular injection
Positive Pregnancy Test Rate | 2 weeks post embryo transfer
Embryo Implantation Rate | 3 weeks post embryo transfer
Clinical Pregnancy Rate | 5 weeks post embryo transfer
Ectopic Pregnancy Rate | 7 weeks' gestation
Ongoing Pregnancy Rate | 10 weeks post embryo transfer
Miscarriage Rate | Prior to 28 weeks' gestation
Drug-Related Venous Thromboembolism (VTE) Rate | Treatment initiation until 10 weeks' gestation
Preterm Birth Rate | 22, 28, 32, 37 weeks' gestation
Gestational Diabetes Mellitus (GDM) Incidence | 24-28 weeks' gestation
Rate of Hypertension in Pregnancy | 20 weeks' gestation to delivery
Low Birth Weight Rate | Delivery
Very Low Birth Weight Rate | Delivery
Macrosomia Rate | Delivery
Extreme Macrosomia Rate | Delivery
Multiple Pregnancy Rate | 6-8 weeks' gestation
Stillbirth Rate | 28 weeks' gestation to delivery
Neonatal Mortality Rate | First 28 days postnatal
Adverse Event Incidence | Enrollment until 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Yanwen Xu, Principal Investigator — Center for Reproductive Medicine, The First Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Reproductive Medical Center, the First Af liated Hospital of Sun Yat-sen University, Zhongshan 2nd Road, Number 1, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol

REFERENCES:
- [Background] Badawy AM, Elnashar AM, Mosbah AA. Aromatase inhibitors or gonadotropin-releasing hormone agonists for the management of uterine adenomyosis: a randomized controlled trial. Acta Obstet Gynecol Scand. 2012 Apr;91(4):489-95. doi: 10.1111/j.1600-0412.2012.01350.x. PMID 22229256
- [Background] Duhan N, Madaan S, Sen J. Role of the aromatase inhibitor letrozole in the management of uterine leiomyomas in premenopausal women. Eur J Obstet Gynecol Reprod Biol. 2013 Dec;171(2):329-32. doi: 10.1016/j.ejogrb.2013.09.010. Epub 2013 Sep 20. PMID 24103533
- [Background] Harmsen MJ, Van den Bosch T, de Leeuw RA, Dueholm M, Exacoustos C, Valentin L, Hehenkamp WJK, Groenman F, De Bruyn C, Rasmussen C, Lazzeri L, Jokubkiene L, Jurkovic D, Naftalin J, Tellum T, Bourne T, Timmerman D, Huirne JAF. Consensus on revised definitions of Morphological Uterus Sonographic Assessment (MUSA) features of adenomyosis: results of modified Delphi procedure. Ultrasound Obstet Gynecol. 2022 Jul;60(1):118-131. doi: 10.1002/uog.24786. PMID 34587658
- [Background] Selntigia A, Molinaro P, Tartaglia S, Pellicer A, Galliano D, Cozzolino M. Adenomyosis: An Update Concerning Diagnosis, Treatment, and Fertility. J Clin Med. 2024 Sep 3;13(17):5224. doi: 10.3390/jcm13175224. PMID 39274438
- [Background] Struble J, Reid S, Bedaiwy MA. Adenomyosis: A Clinical Review of a Challenging Gynecologic Condition. J Minim Invasive Gynecol. 2016 Feb 1;23(2):164-85. doi: 10.1016/j.jmig.2015.09.018. Epub 2015 Sep 30. PMID 26427702